CLINICAL TRIAL: NCT01461148
Title: Phase I/IIa Study of Immunization With Frameshift Peptides Administered With Montanide® ISA-51 VG in Patients With Advanced MSI-H Colorectal Cancer
Brief Title: Vaccination Against MSI Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oryx GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MicOryx
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
Keywords: UICC stage III/IV MSI-H colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FSP peptides (Experimental): Vaccination with three FSP peptides
  Interventions: Biological: FSP peptides

INTERVENTIONS:
Biological: FSP peptides — 100 ug of each FSP (TAF1B(-1), HT001(-1) and AIM2(-1), weekly for 4 consecutive weeks and repeated every four weeks up to a total of 3 cycles.

SUMMARY:
Patients with advanced microsatellite unstable (MSI-H) colorectal cancer will be vaccinated with three so called frame shift peptides (FSPs), AIM2(-1), HT001(-1) and TAF1B(-1) combined with Montanide® ISA-51 VG. By this, an immune response directed against MSI-induced FSPs that are shared by the majority of MSI-H colorectal cancers can be induced. The aim is to show that vaccination against MSI-induced FSPs is safe and can induce or enhance immune responses against MSI-H colorectal cancer-associated antigens.

DETAILED DESCRIPTION:
The present study is initiated to evaluate vaccination with MSI-specific FSPs in patients with MSI-H colorectal cancer. Specifically, the present study aims at the following questions:

* Evaluation of potential toxicity of the FSP AIM2(-1), HT001(-1), TAF1B(-1)
* Evaluation of the immune response in patients with advanced MSI-H colorectal cancer before vaccination and after vaccination with the FSP AIM2(-1), HT001(-1), TAF1B(-1)

In this context, the present study shall demonstrate whether application of FSP in a vaccination approach is associated with the induction of peptide-related toxicity. Hence, the study marks the first step towards the application of FSP in humans, as it provides information on the safety of FSP as vaccination agents for the first time. Moreover, the study shall provide initial information, whether vaccination with FSP can induce FSP-specific immune responses in patients with MSI-H colorectal cancer. Thus, it shall provide information, whether FSPs AIM2(-1), HT001(-1), and TAF1B(-1) have the potential to elicit peptide-specific immune responses and therefore represent suitable targets for the induction of tumor antigen-specific immune responses in patients with MSI-H tumors.

The present study marks an important milestone towards a potential application of MSI-specific FSP as therapeutic agents in the management of patients with MSI-H tumors, particularly patients with MSI-H colorectal cancer. Long-term goal of this approach is to develop novel tools for (1) the palliative and/or adjuvant therapy of patients with advanced MSI-H colorectal cancer and (2) the preventive application of FSPs in mutation carriers of the HNPCC/Lynch syndrome.

ELIGIBILITY:
Inclusion Criteria:

Phase I part inclusion criteria (inclusion criteria for phase IIa part will be defined later using a study amendment):

* Histologically confirmed, surgically resected colorectal cancer of advanced stage (UICC stage III/UICC stage IV). This comprises patients with lymph node metastases (UICC stage III), metastasis to one distant organ (UICC IV, M1a), to more than one distant organ, or patients with peritoneal carcinosis (UICC IV, M1b)
* Detection of high level microsatellite instability (MSI-H) in the resected tumor sample according to the international consensus criteria (multiplex PCR of quasi-monomorphic microsatellite markers BAT25, BAT26, CAT25), see Appendix 1.
* Prior adjuvant standard therapy (chemotherapy with 5-fluorouracil/folinic acid, oxaliplatin, irinotecan or combinations of these) OR Prior palliative standard therapy in the first, second and third line (chemotherapy with 5-fluorouracil, oxaliplatin, irinotecan or combinations of these and/or treatment with anti-EGFR antibodies cetuximab or panitumumab alone or in combination with chemotherapy) with either complete or partial remission, stable disease, or disease progression under therapy; OR Patient has refused adjuvant or palliative standard therapy (chemotherapy using 5-fluorouracil, oxaliplatin, or regimens combining these).
* Expected survival of at least six months.
* Full recovery from surgery or radiation therapy
* ECOG performance status 0, 1 or 2.
* The following laboratory results:
* Neutrophil count ≥ 1.5 x 109/L
* Lymphocyte count ≥ 0.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Serum bilirubin < 2mg/dL
* Male or female patients ≥ 18 years old
* Last therapy discontinued at least 4 weeks prior to vaccination.
* Patient´s written informed consent for participation in the trial

Exclusion Criteria:

* Prior treatment with FSPs AIM2(-1), HT001(-1) and TAF1B(-1)
* Clinically significant heart disease (NYHA Class IV).
* Other serious illnesses, eg, serious infections requiring antibiotics or bleeding disorders.
* History of immunodeficiency disease or autoimmune disease.
* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available.
* HBV, HCV or HIV positivity.
* Chemotherapy, any type of radiation therapy, or immunotherapy within 4 weeks before study entry
* Concomitant treatment with steroids, antihistaminic drugs, or nonsteroidal anti-inflammatory drugs (unless used in low doses for prevention of an acute cardiovascular event or for pain control). Topical or inhalational steroids are permitted.
* Participation in any other clinical trial
* Pregnancy or lactation.
* Women of childbearing potential who are not using a medically acceptable means of contraception.
* Psychiatric or addictive disorders that may compromise the ability to give informed consent.
* Lack of availability of a patient for immunological and clinical follow-up assessment.
* Brain metastases (symptomatic and non-symptomatic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
immune response against FSP peptides | every two weeks
  A positive immune response is defined as positive delayed-type hypersensitivity (DTH) response against at least one of the peptides or a humoral (ELISA for the detection of FSP-specific IgG/IgM/IgA) and/or CD8 and/or CD4 cellular (IFN gamma ELISpot for the detection of FSP-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against at least one of the three peptides

SECONDARY OUTCOMES:
Tumor response | every 8 weeks
  Tumor response is assessed by CT or MRI scans according to RECIST.
safety | up to 8 months
  Safety as assessed by number and severity of adverse events categorized according to CTC criteria v4.0 and the probability of the induction of immune tolerance. Immune tolerance is defined as significant and sustained decline of antigen-specific cellular immune responses after vaccination compared to the antigen-specific cellular immune response measured before vaccination , as assessed by Interferon-gamma (IFN-g) ELISpot using assay-specific cut-off values.

CONTACTS AND LOCATIONS:
Overall Officials: Elke Jäger, Prof. Dr., Principal Investigator — Krankenhaus Nordwest Frankfurt
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Kloor M, Reuschenbach M, Pauligk C, Karbach J, Rafiyan MR, Al-Batran SE, Tariverdian M, Jager E, von Knebel Doeberitz M. A Frameshift Peptide Neoantigen-Based Vaccine for Mismatch Repair-Deficient Cancers: A Phase I/IIa Clinical Trial. Clin Cancer Res. 2020 Sep 1;26(17):4503-4510. doi: 10.1158/1078-0432.CCR-19-3517. Epub 2020 Jun 15. PMID 32540851
- [Derived] Reuschenbach M, Dorre J, Waterboer T, Kopitz J, Schneider M, Hoogerbrugge N, Jager E, Kloor M, von Knebel Doeberitz M. A multiplex method for the detection of serum antibodies against in silico-predicted tumor antigens. Cancer Immunol Immunother. 2014 Dec;63(12):1251-9. doi: 10.1007/s00262-014-1595-y. Epub 2014 Aug 21. PMID 25143232
- See also: trial background information — http://www.ikf-nordwest.de/fuer-aerzte.html?study=29